CLINICAL TRIAL: NCT07184775
Title: Maternal Continuous Glucose Monitoring Surveillance Compared to Finger-stick Glucose Monitoring in Pregnancies With Type 2 Pregestational Diabetes
Brief Title: CGM Adherence Compared to Finger-stick Glucose Monitoring in Pregnancies With Type 2 Pregestational Diabetes
Acronym: PRECIOUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Huda Al-Kouatly, Associate Professor, Maternal-Fetal Medicine, Medical Genetics and Genomics, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2024-1410
Record Dates: First submitted 2025-09-04; First posted 2025-09-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Pregnancy; Continuous Glucose Monitoring System
Keywords: Type 2 Diabetes; Diabetes; continuous glucose monitor; CGM; adherence; pregnancy; maternal health; prenatal care; glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Continuous glucose monitoring (Active Comparator): Patients in this arm of the study will use a continuous glucose monitoring device for glucose monitoring throughout their pregnancy, linked with a HIPAA-compliant digital application that will document measurements.
  Interventions: Device: Continuous glucose monitor
- Finger stick blood glucose monitoring (Active Comparator): Patients randomized to this arm will perform finger stick blood glucose measurements 4x daily (fasting and 2 hours after each meal) and document their measurements in a glucose log.
  Interventions: Device: Glucometer

INTERVENTIONS:
Device: Continuous glucose monitor — Continuous glucose monitors are sensors that detect interstitial blood glucose measurements and relay values from their sensor to a receiver (typically a cell phone) to document values every 5 minutes.
  Other Names: CGM
  Arms: Continuous glucose monitoring
Device: Glucometer — Glucometer measurement involves a patient performing a finger stick with a lancet to draw blood. They then apply blood to a test strip which is analyzed by a glucometer. The glucose measurement provided by the glucometer is then recorded by the patient in a glucose log.
  Arms: Finger stick blood glucose monitoring

SUMMARY:
The purpose of this study is to compare patient adherence to blood sugar monitoring during pregnancy using two different measurement methods in pregnancies complicated by pregestational type 2 diabetes (T2DM). Pregnant patients with T2DM are at risk of having larger babies, babies with low sugar levels in the first 24 hours of life, higher rates of cesarean delivery, stillbirth (death of baby inside the womb), and hypertensive or high blood pressure disorders of pregnancy, such as preeclampsia. Prior studies have shown that treating high blood sugars in pregnancy with medications can reduce these risks. To determine the amount of medication needed, recording of blood sugar levels is necessary. This trial aims to determine whether continuous blood sugar monitors have improved patient recording of blood sugar levels over finger stick blood sugar measurements.

Patients involved in the study will be assigned to either:

1. Fingerstick glucose monitoring (FSG)
2. Continuous glucose monitoring (CGM)

Patients will be randomize in a 1:1 ratio.

FSG Group: blood sugar is tested four times daily - once fasting and two hours after every meal (post-prandial). Blood will be tested using a glucometer, and values will be recorded in a blood sugar log from the time of enrollment to the time of delivery.

CGM Group: A CGM sensor will be placed on the patient's arm for blood sugar collection every 3-5 minutes. This data is sent to a phone application from the time of enrollment to the time of delivery. These sensors will need to be replaced every 14 days.

Percent adherence will be recorded from the time you were randomized to a study group until delivery.

DETAILED DESCRIPTION:
About 1-2% of pregnant patients in the United States have pregestational type 2 diabetes (T2DM). The current standard of care for patients needing pharmacotherapy is to initiate basal and postprandial insulin as determined by the patient's reported blood glucose levels after a week of finger-stick glucose monitoring (FSG). This approach is dependent on the patient performing four finger sticks daily and keeping a record of those values. Titration of medication is also dependent on this process. Patient adherence with finger stick glucose testing is reported at about 50%. Continuous glucose monitors (CGMs) allow for continuous collection of blood glucose data without the patient needing to stick themselves or record their values. Increased adherence has been associated with improved maternal and neonatal outcomes. The goal of this randomized control trial is to determine if CGMs have greater adherence compared to FSG.

The investigator's first aim is to compare adherence to glucose monitoring using CGM versus finger stick monitoring in pregnant patients with T2DM. The investigator's second aim is to compare neonatal and maternal outcomes using CGM versus finger stick monitoring in pregnant patients with T2DM. The investigators hypothesize that CGMs will have increased adherence compared to finger stick glucose monitoring. The investigators also hypothesize that CGM will lead to improved glycemic control, improved neonatal outcomes, and improved maternal outcomes compared to finger stick glucose monitoring.

This is a prospective randomized controlled trial (RCT) comparing adherence to CGM versus FSG in patients with pregestational T2DM prior to initiating prenatal care. T2DM will be defined as the American Diabetes Association (ADA) criteria for diagnosis prior to the date of conception. Patients will receive a CGM after diagnosis will target blood glucose ranges between 65-140 mg/dL.

Participants will be screened, consented, and recruited at their initial prenatal visit. They will then be randomized to either the control FSG arm or the intervention CGM arm. Patients with T2DM are seen every 1 to 2 weeks for medication titration and BG checks, and the investigators would continue this workflow, following patients to delivery. If the patient requires insulin uptitration, a weight-based regimen as described by the ADA will be used. Patients will be seen every 1-2 weeks to titrate insulin to meet target ranges. The only difference in management between two groups will be the way the investigators measure blood glucose. Any indications for delivery will be managed in the same manner independent of group assignment based on the institution's clinical guidelines. After delivery, the investigators would review the documented neonatal and maternal outcomes and documented adherence.

The primary outcome is percent adherence, which will be calculated as number of days used with >75% of time coverage divided by the number of days from initiation to delivery for CGM and number of values reported divided by 28 (4 values are intended to be reported daily), divided by weeks from initiation to delivery for FSG. Secondary outcome is a composite of adverse neonatal outcomes, including the following measures: stillbirth, miscarriage, large for gestational age (LGA) of neonate defined as birth weight >90th percentile for gestational age, fetal hypoglycemia defined as glucose <40 mg/dL <48 hours after birth or glucose, hyperbilirubinemia, stillbirth or neonatal death, or birth trauma. Another secondary outcome is a composite of adverse maternal outcomes, including the following measures: maternal hypoglycemia < 60 mg/dL, shoulder dystocia, OASIS Injuries, operative delivery or c-section, postpartum hemorrhage, or hypertensive disorder of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* fetuses without anomalies
* diagnosis of Type 2 diabetes
* initiation of prenatal care at <20 weeks gestation

Exclusion Criteria:

* diagnosis of Type 1 diabetes
* allergy to insulin
* inability to wear a continuous glucose monitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Patient glucose monitoring adherence | through pregnancy episode, typically 20-35 weeks
  Compare adherence to glucose monitoring using continuous glucose monitoring versus finger stick monitoring in pregnant patients with Type 2 Diabetes

SECONDARY OUTCOMES:
Fetal/neonatal outcomes | through pregnancy episode, typically 20-35 weeks
  Evaluate differences in fetal/neonatal composite morbidity or mortality between groups, including the following measures: stillbirth, miscarriage, large for gestational age (LGA) of neonate defined as birth weight >90th percentile for gestational age, fetal hypoglycemia defined as glucose <40 mg/dL <48 hours after birth or glucose, hyperbilirubinemia, stillbirth or neonatal death, or birth trauma.
Maternal outcomes | through pregnancy episode, typically 20-35 weeks
  Determine rates of composite maternal severe morbidity or mortality between groups, including the following measures: maternal hypoglycemia < 60 mg/dL, shoulder dystocia, OASIS Injuries, operative delivery or cesarean section, postpartum hemorrhage, or hypertensive disorder of pregnancy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Jefferson Health New Jersey, Sewell, New Jersey
  - Thomas Jefferson University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murphy HR, Rayman G, Lewis K, Kelly S, Johal B, Duffield K, Fowler D, Campbell PJ, Temple RC. Effectiveness of continuous glucose monitoring in pregnant women with diabetes: randomised clinical trial. BMJ. 2008 Sep 25;337:a1680. doi: 10.1136/bmj.a1680. PMID 18818254
- [Background] Wernimont SA, Sheng JS, Tymkowicz A, Fleener DK, Summers KM, Syrop CH, Andrews JI. Adherence to self-glucose monitoring recommendations and perinatal outcomes in pregnancies complicated by diabetes mellitus. Am J Obstet Gynecol MFM. 2019 Aug;1(3):100031. doi: 10.1016/j.ajogmf.2019.100031. Epub 2019 Aug 5. PMID 33345801

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT07184775/Prot_SAP_000.pdf